CLINICAL TRIAL: NCT05188937
Title: Validity and Reliability of the Dual-task Questionnaire in Multiple Sclerosis Patients
Brief Title: Validity and Reliability of the Dual-task Questionnaire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sefa Eldemir, Research Assistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1- MS-DTQ-VALİDİTY
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Dual-Task; Validity; Reliability
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- validity and reliability of Dual-task Questionnaire (Experimental): This study was conducted as "test-retest" design and the psychometric properties of Dual-task Questionnaire were examined in patients with MS.
  Interventions: Procedure: validity and reliability study

INTERVENTIONS:
Procedure: validity and reliability study — Validity and reliability assessment of the Dual-task Questionnaire

SUMMARY:
It is important to increase the independence of Multiple Sclerosis (MS) patients in activities of daily living. Almost all activities of daily living require managing many activities at the same time. For example, walking or standing while talking on the phone. There is a need for easily applicable, reliable and valid scales to evaluate dual-task performance in MS patients. Therefore, the aim of this study is to establish the Turkish cultural adaptation, validity and reliability of the Dual-Task Questionnaire scale in MS patients. This study included a total of 50 patients with MS [age (18-65) years]. Dual-task Questionnaire (DTQ), Timed Up and Go test (TUG) with dual-task and Nine Hole Peg test (9-HPT) with dual-task were applied to the patients. The second evaluation (retest) was carried out by the same physiotherapist one week following the first evaluation (test) in order to measure test-retest reliability.

DETAILED DESCRIPTION:
This study included patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS). DTQ was used to assess the frequency of difficulties associated with daily tasks involving the dual-task. Additionally TUG with dual-task and 9-HPT with dual-task were applied to the patients. An experienced physiotherapist applied all these tests. In order to measure test-retest reliability, a retest was carried out by the same physiotherapist one week following the first evaluation. The construct validity of DTQ was tested by Pearson's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multiple Sclerosis
* Must be able to ambulatory status (Expanded Disability Status Scale score ≤ 6 )
* No relapse in the last 3 mounts

Exclusion Criteria:

* Orthopedic problems
* Visual, perception, and hearing problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Validity and reliability of Dual-Task Questionnaire in patients with MS | one week
  Validity and reliability

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Evans JJ, Greenfield E, Wilson BA, Bateman A. Walking and talking therapy: improving cognitive-motor dual-tasking in neurological illness. J Int Neuropsychol Soc. 2009 Jan;15(1):112-20. doi: 10.1017/S1355617708090152. PMID 19128534